CLINICAL TRIAL: NCT04672408
Title: His Bundle Pacing Versus Right Ventricular Pacing: a Randomized Crossover Study (His-PACE)
Brief Title: His Bundle Pacing Versus Right Ventricular Pacing
Acronym: His-PACE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment since the advent of left bundle branch area pacing
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Haran Burri, MD, Professor, University Hospital, Geneva
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CER_GVA_2021
Record Dates: First submitted 2020-11-28; First posted 2020-12-17 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Pacing-Induced Cardiomyopathy
Keywords: His bundle pacing; Right ventricular pacing; Left ventricular systolic function

STUDY DESIGN:
Intervention Model Description: Randomized crossover double-blind
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- His bundle pacing (Active Comparator): Pacing programmed from the His bundle lead
  Interventions: Device: His bundle pacing
- Right ventricular pacing (Placebo Comparator): Pacing programmed from the right ventricular lead
  Interventions: Device: Right ventricular pacing

INTERVENTIONS:
Device: His bundle pacing — Pacing with capture of the His bundle
  Arms: His bundle pacing
Device: Right ventricular pacing — Pacing from the right ventricular lead (septal or apical)
  Arms: Right ventricular pacing

SUMMARY:
This study will randomize cross-over periods of 6 months of right ventricular pacing and His bundle pacing in patients with baseline left ventricular ejection fraction (LVEF)>40%. The primary outcome measure is LVEF.

DETAILED DESCRIPTION:
Monocentric, randomized, double-blind comparative crossover clinical study.

Patients with a standard pacing indication with >20% ventricular pacing, with a baseline LVEF >40%, implanted with a functioning His bundle lead and a backup right ventricular lead, will be randomized to 6-months periods of right ventricular pacing and of His bundle pacing. The primary outcome is LVEF assessed by gated Equilibrium Radionuclide Angiography. Secondary outcomes are diastolic function, New York Heart Association (NYHA) functional class, quality of life, 6-minute walk test, heart failure hospitalisations and device electrical parameters.

ELIGIBILITY:
Inclusion Criteria:

* Baseline LVEF>40%
* Standard pacing indication with >20% VP
* Functional His bundle lead with confirmed His capture
* Functional right ventricular lead with myocardial capture

Exclusion Criteria:

* Unable to sign an informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Left ventricular ejection fraction | 6 months
  Assessed by gated Equilibrium Radionuclide Angiography

SECONDARY OUTCOMES:
Left ventricular peak filling rate (EDV/s) | 6 months
  Assessed by gated Equilibrium Radionuclide Angiography
NYHA functional class | 6 months
  Investigator evaluation
6-minute walk test | 6 months
  Investigator evaluation
Quality of life measure by SF-36 questionnaire | 6 months
  SF-36 questionnaire; 0-100 score (the higher the score, the better the quality of life)
Right ventricular ejection fraction | 6 months
  Assessed by gated Equilibrium Radionuclide Angiography
Hospital admission for cardiovascular causes | 6 months
  Number of days of admissions for cardiovascular causes
Hospital admission for cardiovascular causes | up to 6 months
  Duration in days of admissions for cardiovascular causes

CONTACTS AND LOCATIONS:
Overall Officials: Haran Burri, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- University Hospital Geneva, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Yareta data repository
Supporting Information: Study Protocol, SAP, CSR
Time Frame: At the ocmpletion of the study
Access Criteria: Open access for at least 15 years (as per Swiss law)